CLINICAL TRIAL: NCT01315847
Title: A Three-Part Positron Emission Tomography Study of Brain CGRP Receptor Occupancy Levels Following Administration of MK-0974, Using [11C]MK-4232 as an Imaging Agent
Brief Title: Positron Emission Tomography (PET) Study of Brain Calcitonin Gene-Related Peptide (CGRP) Receptor Occupancy After Telcagepant Administration (MK-0974-067)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0974-067
Record Dates: First submitted 2011-02-22; First posted 2011-03-15 (Estimated); Results first posted 2014-10-24 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — telcagepant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Participants (Part I) (Experimental): Baseline PET imaging of the brain using [11C]MK-4232 tracer (~300 megabecquerel [MBq]) was performed in healthy participants; this PET data served as the baseline for both Period 1 and 2 of Part I. Subsequently in study Part I, Period 1 the healthy participants received a single 1120 mg dose of telcagepant followed by PET imaging of brain with [11C]MK-4232 tracer (~300 MBq) beginning ~3 hours post telcagepant dose. In Part I, Period 2 the healthy participants received a single 140 mg dose of telcagepant followed by PET imaging of brain with [11C]MK-4232 tracer (~300 MBq) beginning ~2 hours post telcagepant dose. Interval between Part I Period 1 and 2 was to be at least 1 week.
  Interventions: Drug: telcagepant; Drug: [11C]MK-4232
- Participants with Migraine (Part III) (Experimental): In study Part III, Period 1 baseline PET imaging of the brain using [11C]MK-4232 tracer (~300 MBq) was performed in participants with migraine during a migraine attack (ictal phase). Later in Part III, Period 1 the participants with an ongoing migraine attack (ictal phase) received a single 140 mg dose of telcagepant followed by PET imaging of brain with [11C]MK-4232 tracer (~300 MBq) beginning ~2 hours post telcagepant dose. In Part III, Period 2 baseline PET imaging of the brain using [11C]MK-4232 tracer (~300 MBq) was performed in participants with migraine, however, without a migraine attack ongoing (interictal phase). Later in Part III, Period 2 participants with migraine without a migraine attack ongoing (interictal phase) received a single 140 mg dose of telcagepant followed by PET imaging of brain with [11C]MK-4232 tracer (~300 MBq) beginning ~2 hours post telcagepant dose. Interval between Part III Period 1 and 2 was to be at least 1 week.
  Interventions: Drug: telcagepant; Drug: [11C]MK-4232

INTERVENTIONS:
Drug: telcagepant — Single oral doses of telcagepant 1120 mg (Part I - Period 1) and 140 mg (Part I - Period 2; Part III - Period 1 and 2)
  Other Names: MK-0974
Drug: [11C]MK-4232 — Single intravenous doses of ~300 MBq [11C]MK-4232 administered as a 5 minute infusion (Part I - Baseline, Period 1 and 2; Part III - Period 1 Baseline and Period 1, and Period 2 Baseline and Period 2)

SUMMARY:
The purpose of this study is to determine the receptor occupancy (RO) associated with telcagepant (MK-0974) administration based on displacement of [11C]MK-4232 from the CGRP receptors in the brain using PET. The study enrolled healthy participants (Part I) and migraine patients (Part III). Due to a protocol amendment, study Part II was not conducted.

DETAILED DESCRIPTION:
For the 1120 mg (i.e., maximal) telcagepant dose, [11C]MK-4232 was administered and PET scan was started ~3 hours post telcagepant to coincide with the Tmax of the 1120 mg dose. For the 140 mg (i.e., therapeutic) telcagepant dose, [11C]MK-4232 was administered and PET scan was started ~2 hours post telcagepant to correspond with the timing of clinical efficacy measurements of telcagepant for migraine treatment in Phase III studies.

ELIGIBILITY:
Inclusion Criteria:

* Participant (Part III only) agrees to use (or have their partner use) a highly effective method of birth control within the projected duration of the study
* Participant has a Body Mass Index (BMI) ≤32 kg/m2 at the prestudy visit
* Participant (Part III only) has had a history of migraine with or without aura >1 year with at least 1 and ≤8 moderate or severe migraine attacks per month in the last 3 months prior to screening
* Participant is judged to be in good health (apart from migraine) based on medical history, physical examination, vital sign measurements, and laboratory safety tests
* Participant has no clinically significant abnormality on electrocardiogram (ECG)
* Participant has been a nonsmoker and/or has not used nicotine or nicotine containing products for at least approximately 6 months
* Participant is willing to comply with the study restrictions and willing to allow the investigators to place an arterial catheter in the radial artery.

Exclusion Criteria:

* Participant is mentally or legally incapacitated, has significant emotional problems at the time of prestudy (screening) visit or expected during the conduct of the study or has a history of a clinically significant psychiatric disorder over the last 5 years (participant with situational depression in the past 6 to 12 months, but not currently, may be enrolled at the discretion of the investigator)
* Participant has a history of any illness that, in the opinion of the study investigator, might confound the results of the study or poses an additional risk to the subject by their participation in the study
* Participant has an estimated creatinine clearance of ≤80 mL/min
* Participant has a history of stroke, chronic seizures, or major neurological disorder
* Participant has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* Participant has a history of neoplastic disease except 1) adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix 2) other malignancies which have been successfully treated ≥10 years prior to the prestudy (screening) visit where, in the judgment of both the investigator and treating physician, appropriate follow-up has revealed no evidence of recurrence from the time of treatment through the time of the prestudy (screening) visit
* For Part III only: Participant is a nursing mother, has difficulty distinguishing his/her migraine attacks from tension or interval headaches, has a history of predominantly mild migraine attacks or migraines usually resolved spontaneously in less than 4 hours, has basilar or hemiplegic migraine headache, has more than 15 headache-days per month or has taken medication for acute headache on more than 10 days per month in any of the 3 months prior to screening, is taking migraine prophylactic medication, was >50 years of at age of migraine onset, has, in the opinion of the investigator, other confounding pain syndromes, psychiatric conditions such as uncontrolled major depression, dementia or significant neurological disorders other than migraine, has liver function tests, specifically alanine aminotransferase (ALT)/aspartate aminotransferase (AST) and Alkaline Phosphatase are above the upper limit of normal at the prestudy (screening) visit or at recheck within 4 weeks prior to Day 1, is taking strong or moderate Cytochrome P450 3A4 (CYP3A4) inhibitors such as Ketoconazole, Diltiazem or Verapamil
* Participant is unable to refrain from or anticipates the use of any medication, including prescription and non-prescription drugs or herbal remedies
* Participant consumes excessive amounts of alcohol
* Participant consumes excessive amounts, defined as greater than 6 servings of caffeinated beverages per day
* Participant has had major surgery, donated or lost 1 unit of blood (approximately 500 mL) or participated in another investigational study within 4 weeks prior to the prestudy visit
* Participant has a history of significant multiple and/or severe allergies (including latex allergy), or has had an anaphylactic reaction or significant intolerability to prescription or non-prescription drugs or food
* Participant is currently a regular user (including "recreational use") of any illicit drugs or has a history of drug (including alcohol) abuse within approximately 2 years
* Participant has participated in a PET study or other study involving administration of a radioactive substance or ionizing radiation within 12 months prior to the prestudy visit
* Participant has implanted or embedded metal objects or fragments in the head or body that would present a risk during the magnetic resonance imaging (MRI) scanning
* Participant suffers from claustrophobia and would be unable to undergo MRI or PET scanning
* Any concern by the investigator regarding the safe participation of the participant in the study, and the ability of the subject to tolerate the procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-01-14 (Actual); Primary Completion 2011-07-26 (Actual); Study Completion 2011-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Hostetler ED, Joshi AD, Sanabria-Bohorquez S, Fan H, Zeng Z, Purcell M, Gantert L, Riffel K, Williams M, O'Malley S, Miller P, Selnick HG, Gallicchio SN, Bell IM, Salvatore CA, Kane SA, Li CC, Hargreaves RJ, de Groot T, Bormans G, Van Hecken A, Derdelinckx I, de Hoon J, Reynders T, Declercq R, De Lepeleire I, Kennedy WP, Blanchard R, Marcantonio EE, Sur C, Cook JJ, Van Laere K, Evelhoch JL. In vivo quantification of calcitonin gene-related peptide receptor occupancy by telcagepant in rhesus monkey and human brain using the positron emission tomography tracer [11C]MK-4232. J Pharmacol Exp Ther. 2013 Nov;347(2):478-86. doi: 10.1124/jpet.113.206458. Epub 2013 Aug 23. PMID 23975906
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0974-067&kw=0974-067&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Due to protocol amendment study Part II was not conducted. One subject who started in Part I, Period 2 had not participated in Part I, Period 1. Therefore, the cumulative total number who started Part I (including those starting in Period 1 and 2) is 6. Study participants were included in either Part I or Part III; none were included in both parts.
Groups:
- Telcagepant and [11C]MK-4232 (Part I): Healthy Participants: Baseline positron emission tomography (PET) imaging of the brain using [11C]MK-4232 tracer (~300 megabecquerel [MBq]) was performed in healthy participants; this PET data served as the baseline for both Period 1 and 2 of Part I. Subsequently in study Part I, Period 1 the healthy participants received a single 1120 mg dose of telcagepant followed by PET imaging of brain with [11C]MK-4232 tracer (~300 MBq) beginning ~3 hours post telcagepant dose. In Part I, Period 2 the healthy participants received a single 140 mg dose of telcagepant followed by PET imaging of brain with [11C]MK-4232 tracer (~300 MBq) beginning ~2 hours post telcagepant dose.
- Telcagepant and [11C]MK-4232 (Part III): Migraineurs: In study Part III, Period 1 baseline PET imaging of the brain using [11C]MK-4232 tracer (~300 MBq) was performed in participants with migraine during a migraine attack (ictal phase). Later in Part III, Period 1 the participants with an ongoing migraine attack (ictal phase) received a single 140 mg dose of telcagepant followed by PET imaging of brain with [11C]MK-4232 tracer (~300 MBq) beginning ~2 hours post telcagepant dose. In Part III, Period 2 baseline PET imaging of the brain using [11C]MK-4232 tracer (~300 MBq) was performed in participants with migraine, however, without a migraine attack ongoing (interictal phase). Later in Part III, Period 2 participants with migraine without a migraine attack ongoing (interictal phase) received a single 140 mg dose of telcagepant followed by PET imaging of brain with [11C]MK-4232 tracer (~300 MBq) beginning ~2 hours post telcagepant dose.
Period: Part I, Period 1
Arm/Group | Telcagepant and [11C]MK-4232 (Part I): Healthy Participants | Telcagepant and [11C]MK-4232 (Part III): Migraineurs
Started | 5 (Subjects who participated in Part I did not participate in Part III.) | 0
Received Telcagepant | 5 | 0
Received [11C]MK-4232 | 5 (One of these participants received [11C]MK-4232 only at baseline.) | 0
Completed | 2 | 0
Not Completed | 3 | 0
Not completed — Reached maximum number of arterial lines | 3 | 0
Period: Part I, Period 2
Arm/Group | Telcagepant and [11C]MK-4232 (Part I): Healthy Participants | Telcagepant and [11C]MK-4232 (Part III): Migraineurs
Started | 3 (One of these subjects did not participate in Part I, Period 1.) | 0
Received Telcagepant | 3 | 0
Received [11C]MK-4232 | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0
Period: Part III, Period 1
Arm/Group | Telcagepant and [11C]MK-4232 (Part I): Healthy Participants | Telcagepant and [11C]MK-4232 (Part III): Migraineurs
Started | 0 | 4 (Subjects who participated in Part III did not participate in Part I.)
Received Telcagepant | 0 | 4
Received [11C]MK-4232 | 0 | 4 (One of these participants received [11C]MK-4232 only at baseline.)
Completed | 0 | 3
Not Completed | 0 | 1
Not completed — [11C]MK-4232 synthesis failure | 0 | 1
Period: Part III, Period 2
Arm/Group | Telcagepant and [11C]MK-4232 (Part I): Healthy Participants | Telcagepant and [11C]MK-4232 (Part III): Migraineurs
Started | 0 | 3
Received Telcagepant | 0 | 3
Received [11C]MK-4232 | 0 | 3
Completed | 0 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study medication (telcagepant and/or [11C]MK-4232).
Groups:
- Telcagepant and [11C]MK-4232 (Part I): Healthy Participants: Baseline PET imaging of the brain using [11C]MK-4232 tracer (~300 MBq) was performed in healthy participants; this PET data served as the baseline for both Period 1 and 2 of Part I. Subsequently in study Part I, Period 1 the healthy participants received a single 1120 mg dose of telcagepant followed by PET imaging of brain with [11C]MK-4232 tracer (~300 MBq) beginning ~3 hours post telcagepant dose. In Part I, Period 2 the healthy participants received a single 140 mg dose of telcagepant followed by PET imaging of brain with [11C]MK-4232 tracer (~300 MBq) beginning ~2 hours post telcagepant dose.
- Total: Total of all reporting groups
Arm/Group | Telcagepant and [11C]MK-4232 (Part I): Healthy Participants | Telcagepant and [11C]MK-4232 (Part III): Migraineurs | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.50 (10.63) | 37.75 (13.20) | 34.60 (11.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4
  Male | 6 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) (Part I)
Description: Any AEs occurring among participants (all were healthy subjects) in Part I of study were recorded. An AE was defined as any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration, whether or not considered related to the study drug. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the administration of the study drug, was also an AE.
Time Frame: Up 14 days after the last dose of telcagepant and/or [11C]MK-4232 in Part I of study (Up to approximately 14 weeks)
Population: All participants who received at least one dose of study medication (telcagepant and/or [11C]MK-4232) in Part I of study.
Measure: Number; unit: participants
Arm/Group | Telcagepant and [11C]MK-4232 (Part I): Healthy Participants
Number analyzed (Participants) | 6
participants | 4

2. Primary Outcome: Number of Participants With AEs (Part III)
Description: Any AEs occurring among participants (all were migraine patients) in Part III of study were recorded. An AE was defined as any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration, whether or not considered related to the study drug. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the administration of the study drug, was also an AE.
Time Frame: Up 14 days after the last dose of telcagepant and/or [11C]MK-4232 in Part III of study (Up to approximately 6 months)
Population: All participants who received at least one dose of study medication (telcagepant and/or [11C]MK-4232) in Part III of study.
Measure: Number; unit: participants
Arm/Group | Telcagepant and [11C]MK-4232 (Part III): Migraineurs
Number analyzed (Participants) | 4
participants | 4

3. Primary Outcome: Brain Calcitonin Gene-related Peptide (CGRP) Receptor Occupancy (RO) Post Telcagepant Obtained by PET Imaging Using [11C]MK-4232 Tracer at Baseline and After a Maximum Dose of Telcagepant (1120 mg) in Healthy Participants (Part I, Period 1)
Description: Brain CGRP RO post telcagepant was determined by change in [11C]MK-4232 PET tracer biokinetics at baseline and post telcagepant administration. Using PET brain images acquired over ~0-90 minutes after [11C]MK-4232 dose, regions of interest (ROIs) were drawn throughout cerebral cortex and white matter, striatum, thalamus, cerebellum and pons. The ROIs were projected onto all frames of the dynamic PET scans in order to generate [11C]MK-4232 tissue time-activity curves (TACs). Serial arterial blood samples for measurement of plasma radioactivity and [11C]MK-4232 concentrations were collected during the PET scans. These samples provided the arterial input function for a two-tissue compartmental model of [11C]MK-4232 tracer biokinetics. Total volume of distribution (VT), an index of receptor density, was estimated by fitting the two-tissue compartmental model to the PET [11C]MK-4232 TACs. Change in VT between baseline and post telcagepant PET studies was used to quantify the brain CGRP RO.
Time Frame: Part I Baseline, at ~0-90 minutes after [11C]MK-4232 dose; and Part I, Period 1 post telcagepant, at ~0-90 minutes after [11C]MK-4232 dose
Population: Participants who received both telcagepant and [11C]MK-4232 during Part I, Period 1 of study, had evaluable data and were compliant with the the study protocol
Measure: Number; unit: percent CGRP RO
Arm/Group | Telcagepant and [11C]MK-4232 (Part I): Healthy Participants
Number analyzed (Participants) | 3
percent CGRP RO
  Subject 04 | 43
  Subject 01 | 48
  Subject 103 | 58

4. Primary Outcome: Average Telcagepant Plasma Concentration During PET Imaging Using [11C]MK-4232 Tracer After a Maximum Dose of Telcagepant (1120 mg) in Healthy Participants (Part I, Period 1)
Description: In Part I, Period 1 blood samples for determination of plasma telcagepant concentrations were obtained prior to the telcagepant dose (time 0) and at 2, 3, 4 and 5 hours post telcagepant dose. The average plasma telcagepant concentration during the PET scan was determined, calculated as the area under the plasma telcagepant concentration versus time curve during the PET scanning interval divided by the duration of the PET scanning interval.
Time Frame: Part I, Period 1 post telcagepant, at ~0-90 minutes after [11C]MK-4232 dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: μM
Arm/Group | Telcagepant and [11C]MK-4232 (Part I): Healthy Participants
Number analyzed (Participants) | 3
μM
  Subject 04 | 16.3 (1.84)
  Subject 01 | 20.2 (3.93)
  Subject 103 | 22.2 (4.43)

5. Primary Outcome: Brain CGRP RO Post Telcagepant Obtained by PET Imaging Using [11C]MK-4232 Tracer at Baseline and After a Therapeutic Dose of Telcagepant (140 mg) in Healthy Participants (Part I, Period 2)
Description: Brain CGRP RO post telcagepant was determined by change in [11C]MK-4232 PET tracer biokinetics at baseline and post telcagepant administration. Using PET brain images acquired over ~0-90 miniutes after [11C]MK-4232 dose, ROIs were drawn throughout the cerebral cortex and white matter, striatum, thalamus, cerebellum and pons. The ROIs were projected onto all frames of the dynamic PET scans in order to generate [11C]MK-4232 tissue TACs. Serial arterial blood samples for measurement of plasma radioactivity and [11C]MK-4232 concentrations were collected during the PET scans. These samples provided the arterial input function for a two-tissue compartmental model of [11C]MK-4232 tracer biokinetics. VT, an index of receptor density, was estimated by fitting the two-tissue compartmental model to the PET [11C]MK-4232 TACs. The change in VT between the baseline and post telcagepant PET studies was used to quantify the brain CGRP RO.
Time Frame: Part I Baseline, at ~0-90 minutes after [11C]MK-4232 dose; and Part I, Period 2 post telcagepant, at ~0-90 minutes after [11C]MK-4232 dose
Population: Participants who received both telcagepant and [11C]MK-4232 during Part I, Period 2 of study, had evaluable data and were compliant with the the study protocol
Measure: Number; unit: percent CGRP RO
Arm/Group | Telcagepant and [11C]MK-4232 (Part I): Healthy Participants
Number analyzed (Participants) | 3
percent CGRP RO
  Subject 02 | 5
  Subject 04 | 10
  Subject 101 | 4

6. Primary Outcome: Average Telcagepant Plasma Concentration During PET Imaging Using [11C]MK-4232 Tracer After a Therapeutic Dose of Telcagepant (140 mg) in Healthy Participants (Part I, Period 2)
Description: In Part I, Period 2 blood samples for determination of plasma telcagepant concentrations were obtained prior to the telcagepant dose (time 0) and at 1, 2, 3 and 4 hours post telcagepant dose. The average plasma telcagepant concentration during the PET scan was determined, calculated as the area under the plasma telcagepant concentration versus time curve during the PET scanning interval divided by the duration of the PET scanning interval.
Time Frame: Part 1, Period 2 post telcagepant, at ~0-90 minutes after [11C]MK-4232 dose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: μM
Arm/Group | Telcagepant and [11C]MK-4232 (Part I): Healthy Participants
Number analyzed (Participants) | 3
μM
  Subject 02 | 0.254 (0.140)
  Subject 04 | 0.859 (0.305)
  Subject 101 | 0.424 (0.187)

7. Primary Outcome: Brain CGRP RO Post Telcagepant Obtained by PET Imaging Using [11C]MK-4232 Tracer at Baseline and After a Therapeutic Dose of Telcagepant (140 mg) in Participants With Migraine During a Migraine Attack (Ictal Phase)(Part III, Period 1)
Description: Brain CGRP RO post telcagepant was determined by change in [11C]MK-4232 PET tracer biokinetics at baseline and post telcagepant administration. Using PET brain images acquired over ~0-90 minutes after [11C]MK-4232 dose, ROIs were drawn throughout the cerebral cortex and white matter, striatum, thalamus, cerebellum and pons. The ROIs were projected onto all frames of the dynamic PET scans in order to generate [11C]MK-4232 tissue TACs. Serial arterial blood samples for measurement of plasma radioactivity and [11C]MK-4232 concentrations were collected during the PET scans. These samples provided the arterial input function for a two-tissue compartmental model of [11C]MK-4232 tracer biokinetics. VT, an index of receptor density, was estimated by fitting the two-tissue compartmental model to the PET [11C]MK-4232 TACs. The change in VT between the baseline and post telcagepant PET studies was used to quantify the brain CGRP RO.
Time Frame: Part III, Period 1 Baseline, at ~0-90 minutes after [11C]MK-4232 dose; and Part III, Period 1 post telcagepant, at ~0-90 minutes after [11C]MK-4232 dose
Population: Results could not be obtained for this measure. For Part III data, the curve fits were unsatisfactory (model curves did not pass through the TAC data points) precluding the quantification of the VT and RO
Arm/Group | Telcagepant and [11C]MK-4232 (Part III): Migraineurs
Number analyzed (Participants) | 0

8. Primary Outcome: Brain CGRP RO Post Telcagepant Obtained by PET Imaging Using [11C]MK-4232 Tracer at Baseline and After a Therapeutic Dose of Telcagepant (140 mg) in Participants With Migraine During Period When Migraine is Absent (Interictal Phase)(Part III, Period 2)
Description: as for outcome 7
Time Frame: Part III, Period 2 Baseline, at ~0-90 minutes after [11C]MK-4232 dose; and Part III, Period 2 post telcagepant, at ~0-90 minutes after [11C]MK-4232 dose
Population: as for outcome 7
Arm/Group | Telcagepant and [11C]MK-4232 (Part III): Migraineurs
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up 14 days after the last dose of telcagepant and/or [11C]MK-4232 (Up to approximately 14 weeks for Part I, Up to approximately 6 months for Part III)
Arm/Group | Telcagepant and [11C]MK-4232 (Part I): Healthy Participants | Telcagepant and [11C]MK-4232 (Part III): Migraineurs
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 4/6 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telcagepant and [11C]MK-4232 (Part I): Healthy Participants (N=6) | Telcagepant and [11C]MK-4232 (Part III): Migraineurs (N=4)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Blood urine present (Investigations) | 0 (0) | 1 (1)
White blood cells urine positive (Investigations) | 0 (0) | 2 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (3)
Migraine (Nervous system disorders) | 0 (0) | 4 (17)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.